CLINICAL TRIAL: NCT03384524
Title: A Phase I/II Evaluation of Bromocriptine, Metoprolol and Tamsulosin Combination Therapy in Eyes With Non-Central Diabetic Macular Edema
Brief Title: Evaluation of Bromocriptine, Metoprolol and Tamsulosin in Eyes With Non-Central DME
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: withdrawn during planning stages
Sponsor: Andrew Moshfeghi, MD, MBA (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Sponsor-Investigator, Andrew Moshfeghi, MD, MBA, Associate Professor of Ophthalmology, Director of Vitreoretinal Surgery Fellowship and Medical Retina Fellowship, Director of Clinical Trials Unit, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: The BEAT DME Study
Record Dates: First submitted 2017-12-15; First posted 2017-12-27 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Bromocriptine; Metoprolol; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combination regiment (Active Comparator): A combination regiment of Bromocriptine (2.5 mg/day), Metoprolol (25 mg/day) and Tamsulosin (0.4 mg/day)
  Interventions: Drug: Bromocriptine 2.5 MG; Drug: Metoprolol 25 MG; Drug: Tamsulosin 0.4 MG
- Placebo (Placebo Comparator): Three placebo pills, matching the external appearance of active drugs
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bromocriptine 2.5 MG — Administered daily
  Other Names: Bromocriptine Mesylate
  Arms: Combination regiment
Drug: Metoprolol 25 MG — Administered daily
  Other Names: Metoprolol Tartrate
  Arms: Combination regiment
Drug: Tamsulosin 0.4 MG — Administered daily
  Other Names: Tamsulosin HCL; Tamsulosin Hydrochloride
  Arms: Combination regiment
Other: Placebo — Three pills, matching active drugs to be administered daily
  Arms: Placebo

SUMMARY:
This phase I/II trial is designed to provide proof of concept evidence that combination therapy can have a beneficial effect on DME and possibly prevent increases in retinal volume or progression of non-central DME into the central subfield of the macula. If a beneficial effect is apparent in this phase I/II study involving a relatively small sample size and short follow-up period, its results could be used to in plan future phase III trials. We believe this study will be the first to show that a systems pharmacology approach can successfully address diabetic macular edema, and thus revolutionize the treatment of complex retinal diseases for which there are a paucity of effective treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Type 1 or type 2 diabetes mellitus
* Best corrected visual acuity using the early treatment diabetic retinopathy study (ETDRS) visual acuity test letter score ≥ 74 (i.e., 20/32 or better) within 30 days of enrollment.
* On clinical exam, definite retinal thickening due to DME within 3,000 μm of the center of the macula but not involving the 500 μm central subfield.
* Thickened non-central macular subfields on the spectral domain OCT macular map
* Central subfield thickness within threshold definition for normal central subfield thickness
* No focal/grid laser within the last 6 months or other treatment for DME within the last 4 months.
* Pseudophakia

Exclusion Criteria:

* Patients with active proliferative diabetic retinopathy
* Pan retinal photocoagulation within the last 12 months of study initiation
* A condition that, in the opinion of the investigator, would preclude participation in the study, e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control.
* Subjects experiencing poor glycemic control who, within the last 4 months, initiated intensive insulin treatment (a pump or multiple daily injections) or plan to do so in the next 4 months.
* Use of systemic corticosteroids or anti-VEGF (vascular endothelial growth factor) therapy.
* Participation in an investigational trial that involves treatment with any drug within 30 days of randomization that has not received regulatory approval at the time of study entry.

Note: study participants cannot receive another investigational drug while participating in this study.

* Known allergy or hypersensitivity to any component of the study drugs.
* Postpartum women with a history of coronary artery disease or other severe cardiovascular conditions (a bromocriptine contraindication).
* Planned glaucoma surgery (floppy iris syndrome associated with tamsulosin therapy).
* Blood pressure > 180/110 mmHg (systolic above 180 or diastolic above 110 mmHg).
* If blood pressure is brought below 180/110 by anti-hypertensive treatment, an individual can become eligible.
* Subjects with second or third degree heart block (metoprolol contraindication).
* Subjects with asthma or other bronchospastic disease (metoprolol precaution).
* Individuals currently taking one of the study medications or a medication in the same therapeutic class (beta receptor antagonists, alpha-1 receptor antagonists, or bromocriptine).
* Participants expecting to move out of the area of the clinical center to an area not covered by another clinical center during the 12 months of the study.
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 12 months. Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment will be used to determine when a pregnancy test is needed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change in retinal volume | 14 months
  Effects of bromocriptine/metoprolol/tamsulosin combination therapy on macular retinal volume compared with placebo in eyes with non-central diabetic macular edema (DME)

SECONDARY OUTCOMES:
Progression of non-central DME compared to central DME | 14 months
  Effects of therapy with bromocriptine/metoprolol/tamsulosin on central subfield thickness and compare the progression of non-central DME to central DME as determined by stereoscopic fundus photographs.
Progression of non-central DME compared to central DME | 14 months
  Effects of therapy with bromocriptine/metoprolol/tamsulosin on central subfield thickness and compare the progression of non-central DME to central DME as determined by Optical Coherence Tomography (OCT).
Change in retinal density | 14 months
  Measured by OCT-angiography
Foveal avascular changes | 14 months
  Measured by fluorescein angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A. Moshfeghi, MD, MBA, Principal Investigator — Associate Professor of Ophthalmology; Director of Vitreoretinal Surgery and Medical Retina Fellowship; Director of Clinical Trials Unit